CLINICAL TRIAL: NCT05844072
Title: The Effect of Mobilization With Movement (MWM) on Weight Bearing Ankle Dorsiflexion (DF) Range of Motion in Individuals With Limited DF Range of Motion
Brief Title: Effect of Mobilization With Movement on Weight Bearing Ankle Dorsiflexion Range of Motion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Cathy Arnot, Principal Investigator, University of South Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00125551
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Ankle Joint Contracture
MeSH Terms: interventions — Movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator setting up the goniometer will be masked to the outcome measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ankle dorsiflexion range of motion with inclinometer in standing (Active Comparator): The Standing Ankle Dorsiflexion Screen (SADS) will be used as a categorical outcome measure which is a more functional way to measure ankle dorsiflexion and does not require the use of additional equipment. The participant will be instructed to stand in tandem stance, one foot directly in front of the other, and bend both knees as far as they can while keeping their heel in contact with the ground. The examiner will then use a ruler to align the posterior knee with the medial malleolus and determine the position of behind, within, or in front of the malleolus.
  Interventions: Procedure: Mobilization with movement
- Weight bearing lunge test (Active Comparator): The Weight Bearing Lunge Test (WBLT) will be used to measure closed chain dorsiflexion in participants. A bubble inclinometer will be placed 15 cm below the tibial tuberosity for measurement during the WBLT. Participants will place their foot on a line on the floor which is perpendicular to the wall to help maintain alignment. The participant's heel will be stabilized by an examiner, and they will then be instructed to lunge forward so that their knee reaches a vertical line on the wall. The measurement will then be taken using the inclinometer placed at 15 cm below the tibial tuberosity. The examiner stabilizing the heel will hold the inclinometer in place, while another examiner ensures proper placement of the inclinometer and takes the reading. The WBLT will be completed twice and the average of the two measurements will be taken.
  Interventions: Procedure: Mobilization with movement

INTERVENTIONS:
Procedure: Mobilization with movement — All participants will receive the MWM intervention with weight bearing ankle dorsiflexion range of motion measured prior to the intervention, immediately following the intervention, and 24 hours (+/- 3 hours) following the intervention. The participant will first place their foot on a 16-inch box to assist in performance of the intervention by the therapist. A licensed physical therapist (PT) will then stabilize the talus for a proper joint mobilization to be performed. The therapist will then mobilize the distal tib/fib in the posterior to anterior direction at end range DF reached through a forward lunge, using a Mulligan's mobilization belt around the distal tibia-fibula. The participant will perform 3 sets of 10 repetitions of the forward lunge and the PT will perform a bout of overpressure at end range during each repetition. Two other investigators will be on either side of participant to assist with balance during the intervention if needed.

SUMMARY:
Limited ankle range of motion is associated with increased risk for ankle sprains, knee joint dysfunction and injury to the ACL. Therefore, it is important that researchers and clinicians understand the best treatment options to increase ankle range of motion for injury prevention. We are recruiting adults with limited ankle range of motion who are lacking current ankle injuries for a treatment investigation. All study procedures will occur on the campus of the University of South Carolina by a licensed Physical Therapist and experienced researcher.

DETAILED DESCRIPTION:
All participants will receive the MWM intervention with weight bearing ankle dorsiflexion range of motion measured prior to the intervention, immediately following the intervention, and 24 hours (+/- 3 hours) following the intervention. The participant will first place their foot on a 16-inch box to assist in performance of the intervention by the therapist. A licensed physical therapist (PT) will then stabilize the talus for a proper joint mobilization to be performed. The therapist will then mobilize the distal tib/fib in the posterior to anterior direction at end range DF reached through a forward lunge, using a Mulligan's mobilization belt around the distal tibia-fibula. The participant will perform 3 sets of 10 repetitions of the forward lunge and the PT will perform a bout of overpressure at end range during each repetition. Two other investigators will be on either side of participant to assist with balance during the intervention if needed.

Weight bearing ankle dorsiflexion range of motion will be measured via a primary and secondary measure. The primary measurement will be use of a bubble inclinometer and the secondary measurement will be the standing ankle dorsiflexion screen (SADS).

ELIGIBILITY:
Inclusion Criteria:

* The sole inclusion criterion will be a limitation in active ankle dorsiflexion range of motion to less than 20 degrees in weight bearing in one or both ankles.

Exclusion Criteria:

* Exclusion criteria include self identified feelings of ankle instability or known diagnosis of chronic ankle instability, dermatologic conditions such as open wounds or impaired sensation which inhibit the ability to use the mobilization strap, and inability to get into the testing position or perform a lunge during the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Dorsiflexion range of motion | Immediately after the intervention
  The measurement will then be taken using the inclinometer placed at 15 cm below the tibial tuberosity. The examiner stabilizing the heel will hold the inclinometer in place, while another examiner ensures proper placement of the inclinometer and takes the reading.
Weight bearing lunge test | Immediatley after intervention
  The Weight Bearing Lunge Test (WBLT) will be used to measure closed chain dorsiflexion in participants. A bubble inclinometer will be placed 15 cm below the tibial tuberosity for measurement during the WBLT. Participants will place their foot on a line on the floor which is perpendicular to the wall to help maintain alignment. The measurement will then be taken using the inclinometer placed at 15 cm below the tibial tuberosity. The examiner stabilizing the heel will hold the inclinometer in place, while another examiner ensures proper placement of the inclinometer and takes the reading. The WBLT will be completed twice and the average of the two measurements will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy F Arnot, DPT, Principal Investigator — University of South Carolina
Locations (1):
- Blatt Physical education Building, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No